CLINICAL TRIAL: NCT06134115
Title: Randomized Double-blinded Multi-center Study of Efficacy and Safety of Lipocet® in Patients With Primary Knee Osteoarthritis Grade 3 - 4
Brief Title: LIKEST Study: Lipocet® in Adults With Primary Knee Osteoarthritis Grade 3-4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanutra S.p.a. (Industry)
Collaborators: NEA Clinical S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIP 02/22
Record Dates: First submitted 2023-10-18; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Primary Knee Osteoarthritis Grade 3 - 4
Keywords: Osteoarthritis; Lipocet
MeSH Terms: conditions — Osteoarthritis | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Lipocet®) (Experimental): Participants received Lipocet® (food supplement) 1 sachet orally once a day for 60 days
  Interventions: Dietary Supplement: Lipocet® (food supplement)
- Control group (Placebo) (Placebo Comparator): Participants received Placebo 1 sachet orally once a day for 60 days
  Interventions: Dietary Supplement: Lipocet Placebo

INTERVENTIONS:
Dietary Supplement: Lipocet® (food supplement) — 1 sachet, 10 ml corresponding to 1500 mg of Cetylated fatty acids
  Arms: Treatment group (Lipocet®)
Dietary Supplement: Lipocet Placebo — Lipocet Placebo matching to Lipocet
  Arms: Control group (Placebo)

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of Lipocet® (food supplement) in patients with primary knee osteoarthritis grade 3 - 4

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will undergo no more than a 1-week screening period to determine eligibility for study entry. Patients that meet inclusion criteria and do not have exclusion criteria will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to Lipocet ® (once a day, 10 ml corresponding to 1500 mg of Cetylated fatty acids) or placebo (once a day, 10 ml) during 60 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Patient Information Sheet and Informed Consent Form
2. Patients with primary osteoarthritis classified according to ACR/EULAR criteria
3. Men or women aged ≥ 40 and ≤80 years
4. A disease severity grade 3 or 4 according to the Kellgren-Lawrence classification:

   * grade 0 (none): definite absence of x-ray changes of osteoarthritis
   * grade 1 (doubtful): doubtful joint space narrowing and possible osteophytic lipping
   * grade 2 (minimal): definite osteophytes and possible joint space narrowing
   * grade 3 (moderate): moderate multiple osteophytes, definite narrowing of joint space and some sclerosis and possible deformity of bone ends
   * grade 4 (severe): large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends
5. Patients who are candidates for knee replacements can be included (this criterion is not mandatory)
6. Patients who mark the pain ≥ 4 cm on a VAS
7. Patients who are willing or able to follow doctor's instructions
8. Patients not participating in other clinical trials within 30 days before the screening
9. Patients who have received sufficient explanation for this clinical trial and agreed to participate

Exclusion Criteria:

1. BMI > 32
2. Systemic inflammatory diseases (e.g. fibromyalgia, etc.)
3. Progressive serious medical conditions (such as cancer, AIDS or end-stage renal disease)
4. Patients with major infections in the observation period
5. Renal diseases (serum creatinine concentration more than 1.2 times the upper limit of the normal range according to the central laboratory definition reference values)
6. Liver dysfunction (serum alanine or aspartate transaminase concentrations more than 1.5 times the upper limit of normal

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Pain on the Visual Analogue Scale (VAS scale) on day 60 | From Baseline to Day 60
  Visual analogue scale (VAS) is a validated questionnaire assessing pain intensity during 60 days of treatment. Possible scores range from 0 cm (no pain) to 10 cm (Pain as bad as it could be). Change = (Day 60 - Baseline Score).
Change From Baseline in Knee Range Of Motion (ROM) on day 60 | From Baseline to Day 60
  Flexion, Extension, External rotation, Internal rotation were measured in degrees. Change = (Day 60 - Baseline Result).
Change From Baseline in WOMAC Total score (Western Ontario and MCMaster Osteoarthritis Index Questionnaire) on day 60 | From Baseline to Day 60
  WOMAC is a validated questionnaire assessing functionality during 60 days of treatment. Possible scores result from 0 to 96 score. Change = (Day 60 - Baseline Score). The WOMAC consists of three subscales: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Higher scores represent worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
The number and % of patients with treatment-emergent adverse events | From Baseline to Day 60
  Incidence and severity of adverse events (AEs) that occurred during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maria Sole Rossato, Study Director — Pharmanutra S.p.a.
Locations (3):
- Georgia (3):
  - LLC "Altra Vita", Tbilisi
  - JSC "Evex Hospitals" (Caraps Medline), Tbilisi
  - LLC "Unica", Tbilisi

IPD SHARING:
Plan to Share IPD: No